CLINICAL TRIAL: NCT02407496
Title: Neurophysiological Attention Test (NAT) for Objective Assessment of Attention Deficit Hyperactivity Disorder (ADHD)
Acronym: NAT-I
Status: Completed | Type: Observational
Sponsor: Think Now Incorporated (Industry)
Collaborators: University of California, Los Angeles (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Gregory Simpson, Ph.D., Chief Scientific Officer, Think Now Incorporated
Other Study IDs: TNI-NAT-1; R43MH099709 (NIH)
Record Dates: First submitted 2015-03-27; First posted 2015-04-03 (Estimated); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ADHD: Adults with Attention Deficit Hyperactivity Disorder (ADHD)
  Interventions: Other: Behavioral assessment and NAT EEG tests
- Control: Healthy individuals without ADHD
  Interventions: Other: Behavioral assessment and NAT EEG tests

INTERVENTIONS:
Other: Behavioral assessment and NAT EEG tests — Individuals in both groups are asked to perform standard behavioral tests and an electroencephalography (EEG) test.

SUMMARY:
The purpose of this study is develop a new assessment tool for Attention Deficit-Hyperactivity Disorder (ADHD) and to then test its validity (i.e. ability to discriminate between individuals with ADHD and healthy controls).

DETAILED DESCRIPTION:
The purpose of this study is to develop a novel approach and software for analyzing electroencephalography (EEG) data to identify biomarkers of ADHD. Then to test the ability of this assessment tool to differentiate between adults with ADHD and healthy controls by comparing the classification accuracy of the metrics from the new tool to the classification accuracy of existing behavioral tests for ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Specific inclusion criteria for ADHD are:

  1. meet established DSM-5 criteria for ADHD predominately inattentive or combined subtype with clinically significant levels of impairment, diagnosed by structured clinical interview, the Mini International Neuropsychiatric Interview, and corroborating information
  2. Clinical Global Impression-Severity (CGI-S) score ≥ 4 for ADHD
  3. no lifetime history of DSM-5 bipolar disorder, psychotic disorder, pervasive developmental disorder, obsessive-compulsive disorder, substance abuse, or substance dependence (except nicotine) as assessed wit the MINI
  4. able in the opinion of the investigator to complete all required study procedures.

Exclusion Criteria:

* Exclusion criteria for both groups are:

  1. History of diagnosis of childhood disorder other than ADHD (e.g. autism, dyslexia)
  2. history of any general medical condition likely to require chronic use of medication with identified CNS effects suspected to alter cognitive performance
  3. history of seizure disorder, brain tumor, other major neurological disorder or head injury resulting in loss of consciousness
  4. serious oxygen deprivation
  5. current psychopathology requiring ongoing treatment with antipsychotic medications, mood stabilizers, benzodiazepines, or anticonvulsants
  6. current untreated psychopathology which is rated to be primary in terms of severity (greater than ADHD severity)
  7. current treatment with guanfacine.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults with Attention Deficit Hyperactivity Disorder (ADHD) from local clinics, clinicians. ADHD community resources in the greater Los Angeles area.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-06; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
NAT Slow Fluctuation Measure | A single measurement is made for each individual at DAY 1 - the time of the brain wave test.
  The NAT EEG test simultaneously generates 2 EEG values and 1 behavioral value that are used together as an assessment metric for ADHD. This is a one-time measure to assess its magnitude in ADHD vs Controls.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory V Simpson, Ph.D., Principal Investigator — Think Now, Inc.; Mark S Cohen, Ph.D., Study Director — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States